CLINICAL TRIAL: NCT01094600
Title: Comparison of Secretin Enhanced MRCP to Endoscopic Pancreatic Function Testing in Diagnosing Exocrine Insufficiency in Patients Who Have Undergone Pancreas Cancer Resection
Brief Title: Comparison of Secretin-enhanced Magnetic Resonance Cholangiopancreatography (S-MRCP) to Endoscopic Pancreatic Function Test (ePFT) in Diagnosing Pancreatic Exocrine Insufficiency
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AAAC7911
Record Dates: First submitted 2010-03-25; First posted 2010-03-29 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; Pancreatic resection; Synthetic human secretin; Secretin-enhanced MRCP; Endoscopic pancreatic function test; Pancreatic exocrine insufficiency
MeSH Terms: conditions — Pancreatic Neoplasms; Exocrine Pancreatic Insufficiency | interventions — Secretin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Secretin (Experimental): Single arm (open label).
  Interventions: Drug: Synthetic Human Secretin

INTERVENTIONS:
Drug: Synthetic Human Secretin — Twelve patients will undergo S-MRCP, at a dose of 0.2 ucg/kg per exam. Secretin, provided by the Repligen Corporation, will be administered by IV bolus injection over 30 seconds followed by a 30 second saline flush. The maximum dose of secretin will be 18.5 ucg.
  Other Names: RG1068

SUMMARY:
The aim of our study is to evaluate S-MRCP, in comparison to direct pancreatic function, to measure pancreatic exocrine function in patients who have symptoms suspicious for insufficiency. We hypothesize that S-MRCP imaging parameters will correlate well with the direct pancreatic exocrine functioning.

DETAILED DESCRIPTION:
Surgical resection offers the only hope of cure for pancreatic adenocarcinoma. While perioperative mortality rates have declined in recent years, pancreatic resection is still associated with significant postoperative malnutrition, maldigestion, and glucose intolerance, mostly as a result of pancreatic insufficiency. Quantifying individual pancreatic function remains a challenge, but is essential in improving the survival and quality of life of pancreatic cancer patients. Secretin-enhanced magnetic resonance cholangiopancreatography (S-MRCP) has recently emerged as a widely-accepted noninvasive technique to assess morphological changes in pancreatic ducts, as well as functional secretory capacity of the gland. The aim of our study is to evaluate S-MRCP as a means to evaluate for pancreatic exocrine insufficiency. This will be a prospective study of twelve patients who have undergone pancreatic resection and who have symptoms of abdominal pain, steatorrhea or weight loss. We will be comparing quantitative parameters of S-MRCP (maximal change in pancreatic duct diameter and volume before and after secretin administration) with endoscopic pancreatic function testing (maximal bicarbonate concentration in duodenal aspirate after secretin administration).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Tissue-confirmed diagnosis of pancreatic adenocarcinoma
* Undergone surgical resection for adenocarcinoma no less than 3 months prior to enrollment
* Report significant abdominal pain/bloating or steatorrhea >3x/week or demonstrate weight loss corresponding to >10% of pre-surgery BMI.
* Scheduled for EGD/EUS to investigate the above clinical indicators.

Exclusion Criteria:

* History of any radiation therapy to the abdomen prior to surgery
* Any contraindication to MRI, including but not limited to implanted metal devices (e.g. pacemaker, berry aneurysm clips, neural stimulator, cochlear implants, or metal in the eye)
* Presence of pancreatic duct stent
* Treatment with an investigational drug within 1 month prior to the day of the study drug administration
* Current enrollment in any other interventional study
* Creatinine greater than 2.0
* Significant liver disease, liver masses, or evidence of portal hypertension
* Pregnancy
* History of sensitivity to secretin
* Unwilling or unable to sign informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Primary outcome: correlation between S-MRCP with ePFT | 30 days
  The primary outcome that we will be measuring will be correlation between duodenal filling on S-MRCP (expressed as percent of duct volume change from baseline and maximal values following secretin administration) with maximal bicarbonate concentration from ePFT.

CONTACTS AND LOCATIONS:
Overall Officials: Harold Frucht, MD, Principal Investigator — Columbia University